CLINICAL TRIAL: NCT03055988
Title: An Exploratory, Randomised, Double-blind, Double-dummy, Active-controlled, Two Period Cross-over Study to Investigate the Effect of 6 Weeks Treatment of Orally Inhaled Tiotropium + Olodaterol Fixed Dose Combination (FDC) Delivered by the Respimat® Inhaler With Fluticasone Propionate + Salmeterol FDC Delivered by the Accuhaler® Inhaler, on Left Ventricular Function and Arterial Stiffness in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Cardiovascular Function in COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.36; 2015-002641-66 (EudraCT Number)
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Results first posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol; Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tiotropium/Olodaterol Fixed Dose Combination (Experimental)
  Interventions: Drug: Tiotropium; Drug: Olodaterol
- Fluticasone Propionate + Salmeterol Fixed Dose Combination (Active Comparator)
  Interventions: Drug: Fluticasone propionate; Drug: Salmeterol

INTERVENTIONS:
Drug: Tiotropium — Fixed Dose Combination
  Other Names: INSPIOLTO, SPIOLTO, STIOLTO, VAHELVA, YANIMO
  Arms: Tiotropium/Olodaterol Fixed Dose Combination
Drug: Olodaterol — Fixed Dose Combination
  Other Names: INSPIOLTO, SPIOLTO, STIOLTO, VAHELVA, YANIMO
  Arms: Tiotropium/Olodaterol Fixed Dose Combination
Drug: Fluticasone propionate — Fixed Dose Combination
  Arms: Fluticasone Propionate + Salmeterol Fixed Dose Combination
Drug: Salmeterol — Fixed Dose Combination
  Arms: Fluticasone Propionate + Salmeterol Fixed Dose Combination

SUMMARY:
The objectives of the study are to explore the effect of treatment with tiotropium + olodaterol fixed dose combination (FDC) compared to fluticasone propionate + salmeterol FDC on:

* reversal of left ventricular diastolic dysfunction assessed with cardiac magnetic resonance (CMR) imaging,
* measures of arterial stiffness assessed by CMR and pulse wave analysis (PWA),
* reduction of hyperinflation assessed with body plethysmography and
* post dose spirometry.

ELIGIBILITY:
Inclusion criteria:

* All patients must sign an informed consent consistent with International Council on Harmonisation - Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial, which includes medication washout and restrictions.
* All patients must have a diagnosis of chronic obstructive pulmonary disease for which they are treated with one or more long-acting inhaled bronchodilators prior to enrolment and must meet the following spirometric criteria:

Patients must have stable airway obstruction with a post-bronchodilator Forced Expiratory Volume in 1st second (FEV1) < 70% of predicted normal calculated with European Coal and Steel Community (ECSC) formulas, and a post-bronchodilator FEV1/Forced Vital Capacity (FVC)< 70% at Visit 1

* Patients with hyperinflation at rest defined as Functional Residual capacity (FRC) > 120 % predicted, with post-bronchodilator reversibility greater than and equal to 7,5 % predicted at Visit 1.
* Male or female patients between 40 and 75 years of age (inclusive) on day of signing informed consent.
* Patients with a smoking history of more than 10 pack years.
* Patients with Modified Medical Research Council (mMRC) Dyspnoea score > 1 at Visit 1.
* Patients must be able to perform technically acceptable pulmonary function tests (spirometry and body plethysmography), Cardiac Magnetic Resonance (CMR), brachial blood pressure measurements with Pulse Wave Analysis (PWA) and other tests during the study period as required in the protocol.
* Patients must be able to inhale medication in a competent manner from the Respimat and Accuhaler inhalers and from a metered dose inhaler (MDI).

Exclusion criteria:

* Patients with a significant disease other than Chronic Obstructive Pulmonary Disease (COPD).
* Patients with a clinically relevant abnormal baseline haematology, blood chemistry, or creatinine.
* Patients with a diagnosis of asthma.
* Patients with a COPD exacerbation in the 6 weeks prior to screening (Visit 1) and patients who experience COPD exacerbation or respiratory tract infection during the washout phase prior to randomisation.
* A history of myocardial infarction, cerebrovascular event or coronary artery intervention other than Coronary Artery Bypass Graft (CABG) within 1 year of screening.
* Abnormal and clinically significant 12-lead Electrocardiogram (ECG).
* Hospitalized for heart failure within the past year. Current severe heart failure (New York Heart Association (NYHA) class IV. Ejection fraction <= 40% from Cardiac Magnetic Resonance (CMR) baseline assessment.
* Patients with systolic blood pressure > 140mmHg and/or diastolic blood pressure > 90mmHg at Visit 1.
* A diagnosis of thyrotoxicosis.
* Known active tuberculosis, cardiac sarcoidosis.
* Any malignancy unless free of disease for at least five years.
* A history of cystic fibrosis.
* Clinically evident bronchiectasis.
* Patients with severe emphysema requiring endobronchial interventions within 6 months prior to screening.
* A history of significant alcohol or drug abuse.
* Patients who have undergone thoracotomy with pulmonary resection.
* Patients being treated with any oral ß-adrenergics.
* Patients being treated with oral corticosteroid medication within 6 weeks prior to Visit 1.
* Patients being prescribed long-term home oxygen treatment.
* Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit or patients who are currently in a pulmonary rehabilitation program.
* Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to screening visit.
* Patients with known hypersensitivity to ß-adrenergics drugs, anticholinergic drugs, fluticasone propionate or to any of the excipients, Benzalkonium chloride (BAC), Disodium edentate (EDTA) or Lactose monohydrate (which contains milk proteins) or any other component of the Respimat® or Accuhaler® delivery systems.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Women of childbearing potential not using highly effective methods of birth control.
* Patients who have previously been enrolled in this study or are currently enrolled in another study.
* Patient who are unable to comply with pulmonary medication restrictions prior to randomisation
* Patients with pacemakers and metal implants (i.e. vascular clips and stents, metal silver in patient's eye) and patients with claustrophobia, due to contraindications for CMR.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (10):
- Germany (10):
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Klinische Forschung Berlin GbR, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Praxis Dr. med. Claus Keller, Frankfurt
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - KLB Gesundheitsforschung Lübeck GmbH, Lübeck
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - RoMed Kliniken, Rosenheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised, double-blind, active-controlled, two-period cross-over study in patients with chronic obstructive pulmonary disease (COPD) to investigate effect of 6-week treatment of tiotropium + olodaterol fixed dose combination (FDC) with fluticasone propionate + salmeterol FDC orally inhaled by the Respimat® and Accuhaler® inhaler respectively.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites which would then ensured that all patients met all inclusion/exclusion criteria. Patients were not to be randomized to trial treatment if any one of the specific entry criteria were not met.
Groups:
- FluticasonePropionate+SalmeterolFDC/ Tiotropium+OlodaterolFDC: Patients orally inhaled total 2 inhalations daily (one inhalation in the morning and evening) via Accuhaler® inhaler of 1000 microgram (μg) fluticasone propionate + 100 μg salmeterol dry powder for inhalation (F+S 1000/100) (500 μg / 50 μg per actuation) for 6-week treatment in period 1 and patients orally inhaled 2 inhalations once daily (in the morning) via Respimat® inhaler of 5 μg tiotropium + 5 μg olodaterol inhalation solution (T+O 5/5) (2.5 μg /2.5 μg per actuation) for 6-weeks treatment in period 2. There was no washout between treatments.
- Tiotropium+OlodaterolFDC/ FluticasonePropionate+SalmeterolFDC: Patients orally inhaled 2 inhalations once daily (in the morning) via Respimat® inhaler of 5 μg tiotropium + 5 μg olodaterol inhalation solution (T+O 5/5) (2.5 μg /2.5 μg per actuation) for 6-week treatment in period 1 and patients orally inhaled total 2 inhalations daily (one inhalation in the morning and evening) via Accuhaler® inhaler of 1000 microgram (μg) fluticasone propionate + 100 μg salmeterol dry powder for inhalation (F+S 1000/100) (500 μg / 50 μg per actuation) for 6-weeks treatment in period 2. There was no washout between treatments.
Period: Period 1
Arm/Group | FluticasonePropionate+SalmeterolFDC/ Tiotropium+OlodaterolFDC | Tiotropium+OlodaterolFDC/ FluticasonePropionate+SalmeterolFDC
Started | 38 | 38
Completed | 37 | 33
Not Completed | 1 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4
Period: Period 2
Arm/Group | FluticasonePropionate+SalmeterolFDC/ Tiotropium+OlodaterolFDC | Tiotropium+OlodaterolFDC/ FluticasonePropionate+SalmeterolFDC
Started | 37 | 33
Completed | 36 | 31
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Other than listed | 1 | 1

BASELINE CHARACTERISTICS:
Population: The treated set (TS): TS is nested within the randomised set and includes all patients who were dispensed study medication and were documented to have taken any dose of study medication. RS includes all patients who signed informed consent form and were also randomised, regardless whether the patient was treated with study medication or not.
Groups:
- Total Patients: Patients orally inhaled total 2 inhalations daily (one inhalation in the morning and evening) via Accuhaler® inhaler of 1000 microgram (μg) fluticasone propionate + 100 μg salmeterol dry powder for inhalation (F+S 1000/100) (500 μg / 50 μg per actuation) or orally inhaled 2 inhalations once daily (in the morning) via Respimat® inhaler of 5 μg tiotropium + 5 μg olodaterol inhalation solution (T+O 5/5) (2.5 μg /2.5 μg per actuation). Patients were randomly assigned to a treatment sequence in two 6-week periods. There was no washout between treatments.
Arm/Group | Total Patients
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.86 (7.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 76
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 75
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular End Diastolic Volume Index (LVEDVI) in the 6th Week of Treatment
Description: LVEDVI is normalised left ventricular end diastolic volume, divided by body surface area.
  Baseline was defined as the value obtained during the assessment performed in a week prior to Visit 2 (Day 1). The change from baseline was calculated as the value obtained in a week prior to Visits 3 and 4 (end of each treatment periods) minus the baseline value.
Time Frame: Baseline and 6 weeks
Population: FullAnalysisSet (FAS)ExcludingExacerbation (FAS-EE) nested within FAS and data from patients who had an exacerbation during treatments were excluded from this set. FAS nested within treated set and included patients who had baseline measurement and at least one post-baseline measurement for primary or secondary endpoints. (Including available data)
Measure: Least Squares Mean (Standard Error); unit: Millilitre/ meter^2 (mL/m^2)
Groups:
- Fluticasone Propionate + Salmeterol FDC (F+S 1000/100): Patients orally inhaled total 2 inhalations daily (one inhalation in the morning and evening) via Accuhaler® inhaler of 1000 microgram (μg) fluticasone propionate + 100 μg salmeterol dry powder for inhalation (F+S 1000/100) (500 μg / 50 μg per actuation) for 6-week treatment period.
- Tiotropium + Olodaterol FDC (T+O 5/5): Patients orally inhaled 2 inhalations once daily (in the morning) via Respimat® inhaler of 5 μg tiotropium + 5 μg olodaterol inhalation solution (T+O 5/5) (2.5 μg /2.5 μg per actuation) for 6-week treatment period.
Arm/Group | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) | Tiotropium + Olodaterol FDC (T+O 5/5)
Number analyzed (Participants) | 59 | 59
Millilitre/ meter^2 (mL/m^2) | 2.855 (1.137) | 2.317 (1.136)
Statistical Analysis 1: Comparison: Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) vs Tiotropium + Olodaterol FDC (T+O 5/5); Mixed model repeated measures (MMRM) model included treatment and period as fixed effects, patient as a random effect and baseline as covariate. Unstructured covariance structure was used for within patient variation. H0: Mean change from baseline in LVEDVI for (Tiotropium + Olodaterol) = Mean change from baseline in LVEDVI for (Fluticasone propionate + Salmeterol); Test type: Superiority; p = 0.6331, Mixed model repeated measures (MMRM); Kenward-Roger approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = -0.537, 95% CI 2-sided [-2.779 to 1.705], Standard Error of Mean 1.120 — Mean difference means the treatment difference vs. F+S (i.e. T+O 5/5 - F+S 1000/100)

2. Secondary Outcome: Change From Baseline in Aortic Distensibility After 6 Weeks of Treatment
Description: Change from baseline in aortic distensibility is presented. Aortic distensibility measurements as measure of arterial stiffness were derived from cine images acquired at end-expiration in planes perpendicular to the thoracic aorta at the level of the pulmonary artery (ascending and descending section of thoracic aorta), abdominal aorta, and perpendicularly to the main, right, and left pulmonary arteries.
Time Frame: Baseline and 6 weeks
Population: FAS-EE set including participants with available data for change from baseline in aortic distensibility.
Measure: Least Squares Mean (Standard Error); unit: Percentage/millimeter of mercury(%/mmHg)
Arm/Group | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) | Tiotropium + Olodaterol FDC (T+O 5/5)
Number analyzed (Participants) | 57 | 57
Percentage/millimeter of mercury(%/mmHg) | -0.006 (0.036) | -0.005 (0.036)
Statistical Analysis 1: Comparison: Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) vs Tiotropium + Olodaterol FDC (T+O 5/5); MMRM model included treatment and period as fixed effects, patient as a random effect and baseline as covariate. Unstructured covariance structure was used for within patient variation; Test type: Superiority; p = 0.9817, Mixed model repeated measures (MMRM); Kenward-Roger approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = 0.001, 95% CI 2-sided [-0.072 to 0.074], Standard Error of Mean 0.036 — Mean difference means the treatment difference vs. F+S (i.e. T+O 5/5 - F+S 1000/100)

3. Secondary Outcome: Change From Baseline in Pulmonary Artery Pulsatility After 6 Weeks of Treatment
Description: Change from baseline in pulmonary artery pulsatility (PAP) is presented. Pulmonary artery pulsatility measurements as measure of arterial stiffness were derived from cine images acquired at end-expiration in planes perpendicular to the thoracic aorta at the level of the pulmonary artery (ascending and descending section of thoracic aorta), abdominal aorta, and perpendicularly to the main, right, and left pulmonary arteries.
Time Frame: Baseline and 6 weeks
Population: FAS-EE set including participants with available data for change from baseline in pulmonary artery pulsatility.
Measure: Least Squares Mean (Standard Error); unit: Percentage of PAP (%)
Arm/Group | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) | Tiotropium + Olodaterol FDC (T+O 5/5)
Number analyzed (Participants) | 57 | 57
Percentage of PAP (%) | -0.175 (1.837) | 1.105 (1.836)
Statistical Analysis 1: Comparison: Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) vs Tiotropium + Olodaterol FDC (T+O 5/5); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5238, Mixed model repeated measures (MMRM); Kenward-Roger approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = 1.280, 95% CI 2-sided [-2.719 to 5.279], Standard Error of Mean 1.995 — Mean difference means the treatment difference vs. F+S (i.e. T+O 5/5 - F+S 1000/100)

4. Secondary Outcome: Change From Baseline in Central Systolic Pressure After 6 Weeks of Treatment
Description: Change from baseline in central systolic pressure is presented.
Time Frame: Baseline and 6 weeks
Population: FAS-EE set including participants with available data for change from baseline in central systolic pressure.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) | Tiotropium + Olodaterol FDC (T+O 5/5)
Number analyzed (Participants) | 58 | 58
mmHg | 0.202 (1.559) | 2.271 (1.559)
Statistical Analysis 1: Comparison: Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) vs Tiotropium + Olodaterol FDC (T+O 5/5); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2687, Mixed model repeated measures (MMRM); Kenward-Roger approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = 2.069, 95% CI 2-sided [-1.640 to 5.779], Standard Error of Mean 1.853 — Mean difference means the treatment difference vs. F+S (i.e. T+O 5/5 - F+S 1000/100)

5. Secondary Outcome: Change From Baseline in Pulse Pressure After 6 Weeks of Treatment
Description: Change from baseline in pulse pressure is presented.
Time Frame: Baseline and 6 weeks
Population: FAS-EE set including participants with available data for change from baseline in pulse pressure.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) | Tiotropium + Olodaterol FDC (T+O 5/5)
Number analyzed (Participants) | 58 | 58
mmHg | 0.170 (1.014) | 0.579 (1.014)
Statistical Analysis 1: Comparison: Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) vs Tiotropium + Olodaterol FDC (T+O 5/5); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7604, Mixed model repeated measures (MMRM); Kenward-Roger approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = 0.409, 95% CI 2-sided [-2.264 to 3.082], Standard Error of Mean 1.335 — Mean difference means the treatment difference vs. F+S (i.e. T+O 5/5 - F+S 1000/100)

6. Secondary Outcome: Change From Baseline in Aortic Augmentation Index After 6 Weeks of Treatment
Description: Change from baseline in aortic augmentation index is presented. Augmentation index was derived from brachial pulse wave separation analysis as augmentation pressure (pressure difference between the reflection wave to the ejection wave) divided by central pulse pressure (at the central aortic site) multiplied by 100.
Time Frame: Baseline and 6 weeks
Population: FAS-EE set including participants with available data for change from baseline in aortic augmentation index.
Measure: Least Squares Mean (Standard Error); unit: Percentage of index (%)
Arm/Group | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) | Tiotropium + Olodaterol FDC (T+O 5/5)
Number analyzed (Participants) | 58 | 58
Percentage of index (%) | 1.723 (1.175) | 1.404 (1.175)
Statistical Analysis 1: Comparison: Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) vs Tiotropium + Olodaterol FDC (T+O 5/5); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8330, Mixed model repeated measures (MMRM); Kenward-Roger approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = -0.320, 95% CI 2-sided [-3.341 to 2.702], Standard Error of Mean 1.509 — Mean difference means the treatment difference vs. F+S (i.e. T+O 5/5 - F+S 1000/100)

7. Secondary Outcome: Change From Baseline in Functional Residual Capacity Body Plethysmography (FRCpleth) % Predicted After 6 Weeks of Treatment
Description: Change from Baseline in Functional Residual Capacity Body Plethysmography (FRCpleth) % predicted is presented. Functional residual capacity, percent predicted is a lung volume at the end of normal expiration assessed/measured by body plethysmography and compared to predicted capacity for such subject, if nonsmoker and without a disease which could compromise their ventilator function, to give a percentage predicted.
Time Frame: Baseline and 6 weeks
Population: FAS-EE set including participants with available data for change from baseline in FRCpleth.
Measure: Least Squares Mean (Standard Error); unit: Percentage of FRCpleth (%)
Arm/Group | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) | Tiotropium + Olodaterol FDC (T+O 5/5)
Number analyzed (Participants) | 59 | 59
Percentage of FRCpleth (%) | -10.211 (2.066) | -18.168 (2.065)
Statistical Analysis 1: Comparison: Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) vs Tiotropium + Olodaterol FDC (T+O 5/5); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0019, Mixed model repeated measures (MMRM); Kenward-Roger approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = -7.957, 95% CI 2-sided [-12.865 to -3.050], Standard Error of Mean 2.452 — Mean difference means the treatment difference vs. F+S (i.e. T+O 5/5 - F+S 1000/100)

8. Secondary Outcome: Change From Baseline in 1.5 Hour Post Dose Forced Expiratory Volume in 1st Second (FEV1) After 6 Weeks of Treatment
Description: Change from baseline in 1.5 hour post dose Forced Expiratory Volume in 1st second (FEV1) is presented.
Time Frame: Baseline and 6 weeks
Population: FAS-EE set including participants with available data for change from baseline in FEV1.
Measure: Least Squares Mean (Standard Error); unit: Litre (L)
Arm/Group | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) | Tiotropium + Olodaterol FDC (T+O 5/5)
Number analyzed (Participants) | 59 | 59
Litre (L) | 0.158 (0.037) | 0.339 (0.037)
Statistical Analysis 1: Comparison: Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) vs Tiotropium + Olodaterol FDC (T+O 5/5); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Mixed model repeated measures (MMRM); Kenward-Roger approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = 0.180, 95% CI 2-sided [0.121 to 0.240], Standard Error of Mean 0.029 — Mean difference means the treatment difference vs. F+S (i.e. T+O 5/5 - F+S 1000/100)

9. Secondary Outcome: Change From Baseline in 1.5 Hour Post Dose Forced Vital Capacity (FVC) After 6 Weeks of Treatment
Description: Change from baseline in 1.5 hour post dose Forced Vital Capacity (FVC) is presented.
Time Frame: Baseline and 6 weeks
Population: FAS-EE set including participants with available data for change from baseline in FVC.
Measure: Least Squares Mean (Standard Error); unit: Litre (L)
Arm/Group | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) | Tiotropium + Olodaterol FDC (T+O 5/5)
Number analyzed (Participants) | 59 | 59
Litre (L) | 0.159 (0.054) | 0.445 (0.054)
Statistical Analysis 1: Comparison: Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) vs Tiotropium + Olodaterol FDC (T+O 5/5); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Mixed model repeated measures (MMRM); Kenward-Roger approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = 0.286, 95% CI 2-sided [0.171 to 0.400], Standard Error of Mean 0.057 — Mean difference means the treatment difference vs. F+S (i.e. T+O 5/5 - F+S 1000/100)

ADVERSE EVENTS:
Time Frame: From first drug administration until 21 days after last drug administration, up to 106 days.
Description: Participant flow is presented by treatment sequence whereas adverse events (AEs) are presented by treatments arms and hence the number of participant differs from the number of participant assigned in participant flow. TS was used for AEs. TS is nested within the randomised set and includes all patients who were dispensed study medication and were documented to have taken any dose of study medication.
Arm/Group | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) | Tiotropium + Olodaterol FDC (T+O 5/5)
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/70 | 2/74
Other Adverse Events (participants affected / at risk) | 7/70 | 13/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) (N=70) | Tiotropium + Olodaterol FDC (T+O 5/5) (N=74)
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Propionate + Salmeterol FDC (F+S 1000/100) (N=70) | Tiotropium + Olodaterol FDC (T+O 5/5) (N=74)
Nasopharyngitis (Infections and infestations) | 2 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03055988/SAP_000.pdf
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03055988/Prot_001.pdf